CLINICAL TRIAL: NCT05067868
Title: A Prospective, Open-label, Multicentre, Interventional, Single-arm, Phase IV Study to Evaluate the Safety and Efficacy of Replagal (Agalsidase Alfa [r-DNA Origin]) in Indian Children and Adults With Fabry Disease
Brief Title: A Study of Replagal in Children and Adults With Fabry Disease in India
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-675-4008; 2022-004233-40 (EudraCT Number)
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Replagal (Experimental): Participants with fabry disease will receive Replagal 0.2 milligram per kilogram (mg/kg) intravenous infusion on Day 1 and every 2 weeks up to Week 51.
  Interventions: Biological: Replagal

INTERVENTIONS:
Biological: Replagal — Participants will receive Replagal 0.2 mg/kg, intravenous infusion at Day 1 and every 2 weeks.
  Other Names: Agalsidase alfa

SUMMARY:
The main aim of this study is to learn more about the safety profile of Replagal.

Participants will receive Replagal every 2 weeks at the clinic for about 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Replagal naïve participants (and who are not part of any other program that allows participant to get access to free enzyme replacement therapy [ERT] at the time of study enrollment and during the study period) of any age with confirmed diagnosis of Fabry disease.
2. Participants who have documented confirmed diagnosis of Fabry disease based on proof of gene mutation: α-galactosidase A gene compatible with Fabry disease and/or a deficiency of α-galactosidase A (less than [<] 4.0 nanomole per milliliter per hour (nmol/mL/hour) in plasma or serum or <8 percent (%) of average mean normal in leukocytes and sequencing of GLA gene for females).
3. Participant must have any clinical manifestations of Fabry disease based on investigator's discretion.
4. Participant/legal authorized representative (LAR)/guardian is able to understand and willing to give written informed consent before performing any study specific procedures and willing to adhere to protocol requirements.
5. Female participants of childbearing potential (example, nonsterilised, premenopausal female participants) must have a documented negative pregnancy test prior to administration of the first dose of Replagal in this study. In addition, all female participants of childbearing potential must use a two medically accepted forms of contraception throughout the study, that is, either a barrier method or hormonal contraceptive with norethindrone and ethinyl estradiol or similar active components.
6. Male participant who is nonsterilised and sexually active with a female partner of childbearing potential agrees to use barrier method of contraception (example, condom with or without spermicide) from signing of informed consent throughout the duration of the study.

Note: Female participants not of childbearing potential defined as those who have been surgically sterilized (hysterectomy, bilateral oophorectomy, or tubal ligation) or who are postmenopausal (example, defined as at least 1 year since last regular menses with an appropriate clinical profile [that is, age appropriate, history of vasomotor symptoms]).

Exclusion Criteria:

1. Participants who have received Replagal.
2. Participants with poorly controlled hypertension as per investigator's discretion.
3. Participants with chronic kidney disease (CKD) with estimated Glomerular Filtration rate less than 15 milliliter per minute (mL/min) /1.73 meter square (m^2) and who had/will have kidney transplantation or are currently on dialysis.
4. Participants with any serious hepatic disorder who had abnormal hepatic function test values at screening (when either alanine aminotransferase [ALT] or aspartate aminotransferase [AST] level exceeded the value three times the upper limit of normal [ULN] and total bilirubin 1.5 times as high as the ULN); and deemed as clinically significant by investigator for hematology and biochemistry. These abnormal laboratory values could be discussed with medical monitor before excluding the participant.
5. If female, the participant is pregnant or lactating or intending to become pregnant before participating in this study, during the study; or intending to donate ova during such time period.
6. Participant/LAR/guardian is unable to understand the nature, scope, and possible consequences of the study.
7. Participant is unable to comply with the protocol, example, uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the investigator.
8. If male, the participant intends to donate sperm during the course of this study.
9. Participants who had participated in any other investigational drug study within the past 4 weeks prior to screening.
10. Any participant deemed as unfit for this trial, as per investigator's clinical judgment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the start of study up to 53 weeks
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical (study) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product, whether or not related to the medicinal (study) product. An SAE is any untoward medical occurrence (whether considered to be related to study product or not) that at any dose results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality or birth defect, an important medical event.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | From the study drug administration up to Week 53
  AE is any unfavorable and unintended sign, symptom, or disease temporally associated with study or use of investigational drug product (IP), whether or not the AE is considered related to IP. TEAEs: AEs occurring or worsening at or after first dose of IP or ongoing at time of enrollment. SAE :untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. Severity: Mild: event that does not generally interfere with usual activities of daily living; Moderate: event that interferes with usual activities of daily living, causing discomfort, permanent risk of harm; Severe: AE that interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Number of Participants With Adverse Drug Reactions (ADRs) Related to Replagal | From the study drug administration up to Week 53
  An ADR is defined as a response to a drug which is noxious and unintended, and which occurs at doses normally used in humans for prophylaxis, diagnosis, or therapy of disease, or for the modification of physiological function. Number of participants with ADRs will be reported.
Number of Participants With Infusion-related Reactions of Replagal | From the study drug administration up to Week 53
  Number of participants with infusion-related reactions of Replagal will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline and at Weeks 13, 27, 39, and 53
  Change in eGRF levels will be assessed from baseline up to week 53.
Number of Participants With Change in Frequency and Regimen of Analgesic use of Replagal for Neuropathic Pain | Baseline up to Week 53
  Participants who are already taking analgesics, any change in frequency and regimen of analgesic use will be monitored throughout the study. Number of participants with change in frequency and regimen of analgesic use of Replagal for neuropathic pain will be reported.
Change From Baseline in Urine Concentration of Globotriaosylceramide (Gb3) | Baseline and at Weeks 13, 27, 39, and 53
  Change from baseline in urine concentration of Gb3 will be assessed.
Change From Baseline in Urine Protein Creatinine Ratio | Baseline and at Weeks 13, 27, 39, and 53
  Urine protein creatinine ratio will be assessed.
Percent Change From Baseline in Left Ventricular Mass Index (LVMI) | Baseline and at Weeks 27 and 53
  The 2-dimensional (2D) echocardiogram will be performed within one month of participant enrolment or at the time of screening, Week 27, and Week 53 and the percent change values from baseline in LVMI (gram per meter square [g/m^2]) will be measured and reported.
Percent Change From Baseline in Left Ventricular Wall Thickness | Baseline and at Weeks 27 and 53
  The 2D echocardiogram will be performed within one month of participant enrolment or at the time of screening, Week 27, and Week 53 and the percent change values from baseline in left ventricular muscular thickness will be measured and reported.
Percent Change From Baseline in Ejection Fraction | Baseline and at Weeks 27 and 53
  The 2D echocardiogram will be performed within one month of participant enrolment or at the time of screening, Week 27, and Week 53 and the percent change values from baseline in ejection fraction will be measured and reported.
Percent Change From Baseline in Quality of Life Based on Questionnaire 36-itme Form Survey (SF-36), Version 2, Acute (Physical and Mental Component Summary Scores) | Baseline and at Weeks 27 and 53
  SF-36 is a generic quality-of-life instrument that has been widely used to assess health-related quality of life (HRQL) of participants. SF-36 consist of 36 items that are aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]). Four domains comprised physical component summary (PCS) score (physical functioning, role-physical, bodily pain, general health) and remaining 4 domains comprised mental component summary (MCS) score (vitality, social functioning, role-emotional, mental health). The scores ranges from 0 to 100. Higher scores indicating better HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- India (3):
  - Institute of Child Health, Kolkata
  - All India Institute of Medical Sciences (AIIMS), New Delhi
  - Sir Gangaram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/615c820deb0e19002afd68b4